CLINICAL TRIAL: NCT07219186
Title: Impacts of AB-free Kava on Mitigating Mobility Loss With Aging: A Pilot Study
Brief Title: Kava Aging and Mobility Study
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202500956
Record Dates: First submitted 2025-10-20; First posted 2025-10-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-08

CONDITIONS: Old Adults; Sleep Quality; Kava; Mobility Impairment; Physical Activity and Stress; Physical Impairment; Sedentary Lifestyle in Patients Over 70
Keywords: AB-free Kava; Old adults; Sleep Difficulties; Mobility Limitations
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Motor Activity; Mobility Limitation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AB-free Kava (Experimental)
  Interventions: Drug: AB-free kava
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AB-free kava — AB-free kava (75mg kavalactones per capsule, for a total of 225 mg/day)
  Arms: AB-free Kava
Other: Placebo — Participants will consume microcrystalline cellulose in capsules identical to AB-free kava, which will be provided by Thorne Research. There are no active ingredients in the placebo capsules.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to learn if AB-free kava works to improve mobility and physical function in older adults with sleep difficulties. It will also learn about the safety of AB-free kava. The main questions it aims to answer are:

* Does AB-free kava improve physical function and/or mobility?
* Does AB-free kava effect sleep, stress, or cellular signaling? Researchers will compare AB-free kava to a placebo (a look-alike substance that contains no drug) to see if AB-free kava works to improve mobility and physical functioning.

DETAILED DESCRIPTION:
This research study is testing whether a specially prepared form of kava, a traditional plant-based supplement, can help improve mobility, sleep, and stress in older adults. Kava has been used safely for centuries in the South Pacific as a natural remedy for relaxation and better sleep, but some modern versions raised safety concerns due to rare liver problems. Researchers have developed a safer version called "AB-free kava," which removes compounds (flavokavains A and B) believed to cause liver issues. Early lab and pilot studies suggest AB-free kava may help improve sleep, reduce stress, decrease inflammation, and support physical activity. This pilot clinical trial will enroll 40 sedentary adults age 70+ who have sleep difficulties. Participants will be randomly assigned to receive either AB-free kava (225 mg/day) or a placebo daily for 8 weeks. The study is double-blind, meaning neither participants nor researchers will know which treatment each person is receiving. Participants will complete visits at the start, midpoint (week 4), and end (week 8) of the study. At each visit, researchers will assess walking ability, grip strength, and sleep quality using wearable activity trackers and validated questionnaires. Blood and hair samples will be collected to measure stress hormones and inflammation. Participants will be screened for eligibility based on age, sleep problems, mobility, and general health. Those with significant health conditions, cognitive impairments, or certain medication use will not be eligible. The study aims to test whether AB-free kava is safe, acceptable, and potentially beneficial for improving sleep and physical function in older adults. If results are promising, this could lead to future larger studies testing AB-free kava as a natural option to support healthy aging.

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years
* 8 ≤ Insomnia severity index (ISI) ≤21
* 4m walking speed <1 m/sec and >0.44 m/sec
* Mild to moderate physical impairment (Short Physical Performance Battery score < 10)
* Sedentary lifestyle (< 150 min per week of moderate intensity physical activity) verified by CHAMPS questionnaire
* Willingness and ability to give informed consent
* Willingness to be randomized to the intervention groups
* Availability for participation through duration of study Exclusion Criteria (General)
* Failure to provide informed consent
* History or clinical manifestation of diabetes, cholelithiasis, liver or renal disease, cancer, or progressive, degenerative neurologic disease (e.g., Parkinson's Disease, multiple sclerosis, ALS)
* Abnormal laboratory markers (e.g., renal or liver abnormalities, elevated potassium levels, or hemoglobin and hematocrit below the lower limit of normal)
* Residence in a Skilled Nursing Facility (SNF); residence in an Assisted Living Facility (ALF) or independent housing is allowed
* Self-reported inability to walk one block
* Significant cognitive impairment, defined as a known diagnosis of dementia or a Mini-Mental Status Exam score < 24
* Severe rheumatologic or orthopedic diseases (e.g., awaiting joint replacement, active inflammatory disease)
* Terminal illness with life expectancy less than 12 months, as determined by a physician
* Severe cardiac disease, including NYHA Class III or IV congestive heart failure, clinically significant aortic stenosis, history of cardiac arrest, use of a cardiac defibrillator, or uncontrolled angina
* Severe pulmonary disease, pneumonitis or interstitial lung disease
* Other significant co-morbid disease (e.g. renal failure on hemodialysis) or severe psychiatric disorder (e.g. bipolar, schizophrenia)
* Current use of antidepressant medications, antipsychotic agents, monoamine oxidase inhibitors, anticholinesterase inhibitors (i.e., Aricept)
* Refuses to reduce alcohol use to 3 or fewer alcoholic drinks per week during the study
* Planning to permanently leave the area in the next year
* Blood pressure readings >180/100 at screening
* Participating in another clinical trial or has received an investigational product within 30 days prior to screening/enrollment.

Exclusion Criteria (AB-free kava-related)

* Regular use of any medications that contain acetaminophen
* Current use of any forms of kava and not willing to stop for a 2-week washout period - dietary supplements or beverages
* Current use of antidepressant medications and antipsychotic agents (including monoamine oxidase inhibitors), or anticholinesterase inhibitors (i.e., Aricept)
* Diagnosed with liver dysfunction or with previous liver diseases during the past five years
* Levels of ALT, AST, ALP or total bilirubin over 3xlimit of normal (ULN) range at prescreen

Temporary Exclusion Criteria

* Acute infection (urinary, respiratory, other) or hospitalization within 1 month
* Myocardial infarction, CABG, or valve replacement within past 6 months
* Pulmonary embolism or deep venous thrombosis within past 6 months
* Stroke, hip fracture, hip or knee replacement, or spinal surgery within past 4 months
* Receiving physical therapy for gait, balance, or other lower extremity training

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
400-meter walk test | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  400-m walk test is a feasible, objective, reliable, well-validated measure to assess mobility and is commonly used in large clinical trials. Participants will be asked to walk 400 m at their usual pace, without overexerting, on a 20-m course for 10 laps (40 m/lap). Participants will be allowed to use a cane, but not a walker, to complete this test.
Short Physical Performance Battery (SPPB) | Obtained at screening, from baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  SPPB will be used to assess physical performance, which is based on a timed 4-m walk, balance and chair stand tests with a range from 0 (worst performers) to 12 (best performers). This scale is reliable and valid for predicting institutionalization, mortality and disability SPPB will be administered by a trained and certified examiner.
Grip Strength | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Grip strength test will be used to measure muscle strength and has been widely used as a general indicator of functional status. Grip strength will be measured using the Jammar dynamometer.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Insomnia Severity Index (ISI) will be used to characterize sleep disturbances and measure the severity of insomnia during the trial.
Pittsburgh Sleep Quality Index (PSQI) | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available) to assess the quality of sleep.
Perceived Stress Scale (PSS) | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Perceived Stress Scale (PSS) is a 10-item scale that will measure the perception of stress. It will be used to assess the levels of stress among subjects during the trial and quantity its levels.
Montgomery Asberg Depression Rating Scale (MADRS) | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Montgomery Asberg Depression Rating Scale (MADRS) is a 10-item clinician rated scale to measure depression. It will be used to monitor subjects for changes in severity of depressive symptoms during the trial.
Hair Cortisol | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  A biomarker used to assess long-term cortisol exposure.
C-reactive protein (CRP) | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  C-reactive protein (CRP) is an acute-phase protein produced by the liver in response to inflammation. It serves as a biomarker of systemic inflammation, with higher levels indicating infection, tissue injury, or chronic inflammatory conditions such as cardiovascular or metabolic disease.
Interleukin-6 (IL-6) | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Interleukin-6 (IL-6) is a cytokine that plays a key role in the body's immune response and inflammation, used as a biomarker for systemic inflammation.
Tumor necrosis factor-alpha (TNF-α) | From baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Tumor necrosis factor-alpha (TNF-α) is a pro-inflammatory cytokine produced primarily by macrophages and other immune cells, used as a biomarker for systemic inflammation.
Total sleep time (TST) | Obtained at screening, from baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Total sleep time (TST) will be calculated using wrist-based actigraphy. TST will include the amount of time spent asleep while in bed, obtained in minutes.
Sleep onset latency (SOL) | Obtained at screening, from baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Sleep onset latency (SOL) will be obtained using wrist-based actigraphy. SOL measures the amount of time it takes to fall asleep after getting into bed, measured in minutes.
Sleep efficiency (SE) | Obtained at screening, from baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Sleep efficiency (SE) will be measured using a wrist-based actigraphy. SE measures the percent of time in sleep that is actually spent asleep, obtained in minutes.
Wake after sleep onset (WASO) | Obtained at screening, from baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Wake after sleep onset (WASO) will be obtained using a wrist-based actigraphy. WASO represents the amount of time awake after initially falling asleep, measured in minutes.
Number of wake bouts | Obtained at screening, from baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Number of wake bouts will be measured using wrist-based actigraphy. Number of wake up bouts represents the number of times woken up during the night.
Sedentary activity (SA) | Obtained at screening, from baseline to 4 weeks, and again to the end of treatment at 8 weeks.
  Sedentary activity (SA) will be measured using wrist-based actigraphy, using wrist cut-points. Counts per minute will be used to quantify time spent in sedentary and non-sedentary styles in older adults

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Institute on Aging University of Florida, Gainesville, Florida
  - Institute on Aging Unversity of Florida, Gainesville, Florida

IPD SHARING:
Plan to Share IPD: Undecided